CLINICAL TRIAL: NCT06883097
Title: Hybrid Trial of a Digital Therapeutic for Smoking Cessation Among Persons Living With HIV
Brief Title: Quitting Matters Human Immunodeficiency Virus Hybrid Trial
Acronym: QMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University at Buffalo (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00112958; 7R01CA285331-02 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Tobacco; Tobacco Abstinence; Smoking Cessation; Smoking Cessation; Tobacco Dependence; Human Immunodeficiency Virus (HIV); Tobacco Dependence Caused by Cigarettes; Cancer Prevention
Keywords: Tobacco; Smoking Cessation; Human immunodeficiency virus (HIV); Tobacco Abstinence; Quit Smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Acquired Immunodeficiency Syndrome | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Learn to Quit - HIV (LTQ-H) App (Experimental): a smoking cessation Digital Therapeutic (DTx) for people with HIV (PWH)
  Interventions: Behavioral: Learn to Quit-HIV (LTQ-H) App
- QuitStart App (Active Comparator): an evidence-based DTx designed for the general population
  Interventions: Behavioral: QuitStart

INTERVENTIONS:
Behavioral: Learn to Quit-HIV (LTQ-H) App — LTQ-H consists of 319 screens divided into: (a) HIV-tailored smoking cessation ACT skills, (b) education about tobacco dependence and treatment (USCPG), and (c) NRT psychoeducation and adherence. Content is gradually presented across 28 modules (14 education and 14 skills) that can be completed in 14 days.
  Other Names: a smoking cessation Digital Therapeutic (DTx)
  Arms: Learn to Quit - HIV (LTQ-H) App
Behavioral: QuitStart — This DTx, QuitGuide was adapted from the National Cancer Institute Smokefree.gov Initiative's QuitGuide's 5 modules have the following intervention components: (a) psychoeducation about the impact of smoking on health, (b) setting up a quit date and a quit plan, (c) selecting reasons for quitting, (d) tracking triggers and smoking habits, and (e) tips for quitting.
  Other Names: an evidence-based DTx designed for the general population
  Arms: QuitStart App

SUMMARY:
The purpose of this study is to compare the advantages and disadvantages of two approaches for quitting smoking among people living with HIV (PWH). Participants will complete a 24- week (~6-month) study where the Participants will be assigned to one of two smartphone apps to help with quitting smoking. Regardless of the group participants are assigned to, they will also receive a combination of nicotine replacement therapy (patches and gums) that have been shown to help people quit smoking. The main questions this study aims to answer are:

Participants will complete 5 video call visits over about 6 months. Participants will install their assigned smoking cessation app onto their phone and will be asked to use the app for the duration of the study along with their provided Nicotine Replacement Therapy (NRT) products. During the study visits, participants will meet with study staff to complete questionnaires and interviews. Participants may be asked to provide breath and saliva samples to measure the level of carbon monoxide and nicotine.

DETAILED DESCRIPTION:
Tobacco use has alarmingly high rates among people with Human Immunodeficiency Virus (HIV) (PWH), 43% compared with 15% in the general population. Due to the development of highly effective treatments for HIV and the resulting increased longevity among PWH, this population now loses more life years to smoking than to HIV infection itself. Novel and effective models to deliver wider reaching smoking cessation interventions for PWH are highly needed and indicated as a priority for National Institute of Health. Digital therapeutics (DTx) may be a novel, scalable, and highly available approach for engaging and treating smoking in this population. However, although DTx for smoking cessation have been shown effective in the general population, no large trial to date has examined the effectiveness of a tailored DTx for smoking cessation in PWH, and no implementation science work has examined barriers and facilitators of implementation of DTx for smoking cessation in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported daily cigarette smoking over the past 30 days
2. Self-reported HIV status
3. Age 18 or older
4. Desire to quit smoking
5. Willing and medically eligible to use NRT
6. Currently receiving HIV care
7. Currently owning an Android or iOS smartphone

Exclusion Criteria:

1. Current acute psychotic episode or unsafe to participate in the study
2. Pregnant or intending to become pregnant in the next 6 months
3. Currently receiving any pharmacological and/or behavioral intervention or counseling for smoking cessation
4. Any medical condition or medication that could compromise subject safety, as determined by the PIs and/or study physician
5. Not able to fluently speak and write in English
6. Hearing, comprehension, visual, speech, or motor limitations that preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Biochemically verified 7-day point prevalence abstinence at 6, 12, 18, and 24-weeks | Weeks 6, 12, 18, and 24
  Abstinence is determined by a self-report of not smoking any cigarettes for greater than or equal to 7 days prior to Weeks 6, 12, 18, and 24 and biochemically verified by an expired carbon monoxide breath test or a cotinine level saliva test at Weeks 6, 12, 18, and 24. Criteria for the bioverification tests to be considered abstinent includes a reading of <6 parts per million using an iCOquit Smokerlyzer carbon monoxide breath test OR a cotinine level of 30 or less ng/ml using an iScreen saliva test.
  If the participant does not meet both criteria of the self report of 7 or more days of abstinence plus a bioverification test below the thresholds listed above, they are not considered abstinent. As per convention, participants are assumed to be smoking if they report smoking at the time-point, cannot be reached to provide data at the time-point, fail to provide a breath sample at the time-point, or provide a breath sample at the time-point that is greater than or equal to 6 ppm.

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence at 6 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 6 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 7 days prior to the timepoint.
Self-reported 7-day point prevalence abstinence at 12 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 12 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 7 days prior to the timepoint.
Self-reported 7-day point prevalence abstinence at 18 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 18 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 7 days prior to the timepoint.
Self-reported 7-day point prevalence abstinence at 24 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 24 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 7 days prior to the timepoint.
Self-reported 30-day point prevalence abstinence at 6 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 6 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days but < 30 days prior to the timepoint.
Self-reported 30-day point prevalence abstinence at 12 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 12 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days prior to the timepoint.
Self-reported 30-day point prevalence abstinence at 18 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 18 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days prior to the timepoint.
Self-reported 30-day point prevalence abstinence at 24 weeks - the percentage of participants who are abstinent from cigarettes at a given point in time | 24 weeks
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days prior to the timepoint.
Change in average number of cigarettes smoked per day | 6 weeks
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Change in average number of cigarettes smoked per day | 12 weeks
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Change in average number of cigarettes smoked per day | 18 weeks
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Change in average number of cigarettes smoked per day | 24 weeks
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Average number of quit attempts | 6 weeks
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking cigarettes at all for 24 hours or more.
Average number of quit attempts | 12 weeks
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking cigarettes at all for 24 hours or more.
Average number of quit attempts | 18 weeks
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking cigarettes at all for 24 hours or more.
Average number of quit attempts | 24 weeks
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking cigarettes at all for 24 hours or more.
Average acceptance of physical smoking cravings | 6 weeks
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average acceptance of physical smoking cravings | 12 weeks
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average acceptance of physical smoking cravings | 18 weeks
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average acceptance of physical smoking cravings | 24 weeks
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average frequency of app use | Weeks 0-24
  Average frequency of app use over the 24-week study period. Measured by average number of app openings.
Average duration of app use | Weeks 0-24
  Average duration of app use over the 24-week study period.
Average number of app modules completed | Weeks 0-24
  Average number of app modules completed over the 24-week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vilardaga Viera, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University, Implementation Science, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No